CLINICAL TRIAL: NCT04474535
Title: Association of β-cell Secretory Status With Early Microvascular and Macrovascular Complications in Patients With Type 1 Diabetes Mellitus
Brief Title: C-peptide Correlation With Microvascular Complications in T1DM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Other Study IDs: T1DM C-peptide
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes; C-peptide; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the presence of residual insulin secretion in patients with DM1 and its correlation with the possible protection against early microvascular and macrovascular complications, emphasizing on the functionality of the myocardium.

DETAILED DESCRIPTION:
The study will include approximately 200 patients, male and female, with DM1 who are being followed in the outpatient diabetic clinic of our hospital.

Each patient will visit the Research Laboratory of the Diabetes Centre of our Department. The visit will take place in the morning in a fasting state of about 12 hours. Demographic data will be recorded along with the patients' habits, lifestyle, current medication and complete medical history of concomitant diseases.

This will be followed by anthropometric measurements (weight, height, BMI) and afterwards blood samples will be taken for the determination of urea, creatinine, glucose, HbA1c and lipids. Part of each blood sample will be collected in tubes containing EDTA to determine fasting c-peptide concentrations. The presence of microalbuminuria will be assessed from a morning urine sample by calculating urinary albumin to creatinine ratio (ACR).

The functionality of the heart's autonomic nervous system will be assessed through the use of heart rate variability (HRV) measurements, using the standard Ewing's tests panel: deep inhalation, standing up and Valsalva's manoeuvre. Changes in blood pressure when changing from the supine to the standing position will also be recorded. Subsequently, the distensibility of the large vessels will be determined, by calculating the conduction velocity of the pulse wave between the carotid and the femoral artery (pulse wave velocity (PWV)).

Finally, a full transthoracic echocardiographic study will be carried out to assess functionality, systolic and diastolic, of the left ventricle (LV).

All data will be recorded in an electronic database for statistical processing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Informed consent form

Exclusion Criteria:

* Known macrovascular complications
* Known serious microvascular complications

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with type 1 diabetes followed in our Diabetes outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
C-peptide concentrations | 1 day
  Concentrations of plasma c-peptide in the fasting condition
Microvascular complications | 1 day
  Presence of microvascular complications
Macrovascular complications | 1 day
  Presence of macrovascular complications

SECONDARY OUTCOMES:
Association between c-peptide and complications | 1 day
  Positive or negative association between c-peptide concentrations and presence of microvascular or macrovascular diabetes complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, Principal Investigator — First Department of Propaedeutic Medicine, University of Athens
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece